CLINICAL TRIAL: NCT06631157
Title: Essential Pro Post-Market Clinical Follow-up Study
Brief Title: Essential Pro Study ( rEPIC04E-HK )
Acronym: rEPIC04E-HK
Status: Recruiting | Type: Observational
Sponsor: Fundación EPIC (Other)
Responsible Party: Sponsor
Other Study IDs: rEPIC04E-HK- Pro Study-HK
Record Dates: First submitted 2024-10-02; First posted 2024-10-08 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Coronary Artery Disease; Ischemic Heart Disease
Keywords: MDR (Medical Device Regulations); PMCF (Post-Market Clinical Follow-up); Paclitaxel eluting coronary balloon dilatation catheter
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Coronary Artery Disease (CAD)
  Interventions: Device: Essential pro

INTERVENTIONS:
Device: Essential pro — Patients in whom treatment with (Essential Pro) has been attempted

SUMMARY:
Single center, prospective, non-randomized, post-market clinical follow-up (PMCF) study to confirm and support the clinical safety and performance of Essential Pro to meet EU Medical Device regulation (MDR) requirements in all the CONSECUTIVE patients treated with Essential Pro.

DETAILED DESCRIPTION:
This study intends to analyze:

* Device effectiveness (in its individual use, technical performance) and procedural effectiveness (technical outcome at the end of lesion treatment with the device under study and any other device being used).
* Device safety (in its individual use, technical performance) and procedural safety (technical outcome at the end of lesion treatment with the device under study and any other device being used).
* Clinical outcomes at the end of the procedure and during the specified follow-up period for each device. The follow-up timeframe is established based on the conditions of use and type of device being used, according to the requirements established by the relevant Notified Body.

ELIGIBILITY:
Inclusion Criteria:

* Patient treated with Essential Pro according to routine hospital practice and following instructions for use
* Informed consent signed

Exclusion Criteria:

* Not meet inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with Essential Pro according to routine hospital practice and following instructions for use
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Safety Endpoint. Freedom from Target Lesion Failure | 12 months
  Freedom from TARGET LESION FAILURE (TLF), composite endpoint of cardiac death, myocardial infarction (MI) and a new Target Lesion Revascularization (TLR). Freedom from TARGET LESION FAILURE (TLF), composite endpoint of cardiac death, myocardial infarction (MI) and a new Target Lesion Revascularization (TLR).

SECONDARY OUTCOMES:
Efficacy Endpoint. Freedom from Target Lesion Failure (TLF) | 12 months
  Freedom from TARGET LESION FAILURE (TLF), composite endpoint of Cardiac death, Myocardial infarction, and new Target Lesion Revascularization (TLR).
Freedom from Balloon rupture | During PCI
  Freedom from Balloon rupture
Freedom from Hypotube rupture | During PCI
  Freedom from Hypotube rupture
Freedom from Complicated withdrawal | During PCI
  Freedom from Complicated withdrawal
Freedom from Coronary perforation | During PCI
  Freedom from Coronary perforation
Freedom from Coronary dissection >C | During PCI
  Freedom from Coronary dissection >C
Freedom from No reflow | During PCI
  Freedom from No reflow
Freedom from Coronary thrombosis | During PCI
  Freedom from Coronary thrombosis

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Margaret Hospital, Lai Chi Kok, Hong Kong

REFERENCES:
- [Background] Gruntzig A. Transluminal dilatation of coronary-artery stenosis. Lancet. 1978 Feb 4;1(8058):263. doi: 10.1016/s0140-6736(78)90500-7. No abstract available. PMID 74678
- [Background] Wu X, Li L, He L. Drug-Coated Balloon versus Drug-Eluting Stent in Patients with Small-Vessel Coronary Artery Disease: A Meta-Analysis of Randomized Controlled Trials. Cardiol Res Pract. 2021 Apr 13;2021:1647635. doi: 10.1155/2021/1647635. eCollection 2021. PMID 33953973